CLINICAL TRIAL: NCT00468273
Title: A Clinical Study of Immune Globulin Intravenous (Human) Omr-IgG-am IGIV in Subjects With Primary Immune Deficiency Diseases
Brief Title: A Clinical Study of Intravenous Immunoglobulin
Acronym: IGIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: FFF Enterprises (Industry)
Collaborators: OMRIX Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GAM-PID-03-US; NCT00468273 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2007-05-01; First posted 2007-05-02 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Immunologic Deficiency Syndromes
Keywords: Deficiency Syndromes, Antibody; Antibody Deficiency Syndrome; Bruton's agammaglobulinemia; Common Variable Immune Deficiency; Hyper IgM syndromes
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Bruton type agammaglobulinemia; Common Variable Immunodeficiency; Hyper-IgM Immunodeficiency Syndrome | interventions — gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravenous Immune Globulin (Experimental): Subjects with primary humoral immunodeficiency
  Interventions: Drug: Immune Globulin Intravenous (Human) Omr-IgG-am IGIV

INTERVENTIONS:
Drug: Immune Globulin Intravenous (Human) Omr-IgG-am IGIV — IGIV infusions of 300-900 mg/kg every 3 or 4 weeks

SUMMARY:
The purpose of this study is to measure the pharmacokinetics, efficacy and safety of Immune Globulin Intravenous (Human) [IGIV], 5% Solution Omr-IgG-am™ in patients with primary immunodeficiency diseases.

DETAILED DESCRIPTION:
This is an open label, single-arm, prospective, multi-center, uncontrolled Phase III clinical study to evaluate the efficacy, pharmacokinetics and safety of Omr-IgG-am™ in patients with primary immunodeficiency diseases.

Approximately 50 subjects will be enrolled for 16 Months:

screening- 1 month treatment-12 months follow-up-3 months

Subjects will be infused every 21 to 28 days according to their previous IVIG treatment schedule. Subjects treated every 28 days will receive 13 study IGIV infusions. Subjects treated every 21 days will receive 17 study IGIV infusions.

We will record the incidence of acute infections, especially acute serious bacterial infections, during the year each subjet is on study.

We will record the incidence of adverse events that occur during each infusion and up to 48 hours after each infusion.

At the time the study is explained to the subjects, each investigator will ask all subjects whose body weight is above 37 kg (or greater as defined by local standards) about their willingness to participate in the pharmacokinetic (PK) portion of the study. This will involve 4 additional visits after the 5th or 6th study IGIV infusion in order to draw blood samples for analysis.

ELIGIBILITY:
The following list is incomplete. A complete list is in the protocol.

Inclusion Criteria:

* Ages 3 to 75 years and weigh at least 27 kg.
* Confirmed clinical diagnosis of a Primary Immune Deficiency disease including hypogammaglobulinemia, preferably with documented antibody deficiency, or agammaglobulinemia.
* Has been receiving licensed IGIV for at least 3 months prior to this study.
* Trough IgG levels, dose of IGIV, and treatment intervals for the last 2 consecutive licensed IGIV treatments must be documented.
* The subject or legal guardian has signed the informed consent form. If appropriate, the subject has signed a child assent form.
* The subject or legal representative has signed the HIPAA declaration.

Exclusion Criteria:

* Subjects with isolated IgG subclass deficiency or specific antibody deficiency without hypogammaglobulinemia will not be eligible.
* The subject has a history of hypersensitivity or persistent or repeated adverse reactions to human immunoglobulin.
* The subject has selective IgA deficiency, history of reaction to products containing IgA, or is known to have antibodies to IgA.
* The subject is currently participating, or has participated within the previous 30 days, in another clinical study of an investigational product or device.
* The subject is pregnant or is nursing. Women of childbearing potential must agree to using a method of contraception.
* The subject has had an acute bacterial infection within 28 days of screening.
* The subject is seropositive for any of the following at screening:
* Antibodies to HIV 1&2
* Antibodies to HCV
* HbsAg
* The subject, at screening, has alanine aminotransferase (ALT) levels greater than 2.5 times the upper limit of normal.
* The subject has severe renal impairment.
* The subject has a history of DVT, thrombotic or thrombic complications of IGIV therapy.
* The subject suffers from any acute or chronic medical condition that, in the opinion of the investigator, may interfere with the conduct of the study.
* The subject has an acquired medical condition known to cause secondary immune deficiency or otherwise increase the subject's risk of infection.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2006-11; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Incidence of acute serious bacterial infections | one year
  Acute serious bacterial infections are defined in The FDA(CBER) Guidance for industry for studies of IGIV to support marketing of IGIV as replacement therapy for primary humoral immunodeficiency (June, 2008).

SECONDARY OUTCOMES:
The number of hospitalizations and days of hospitalization per subject per year for PID related infections | during treatment with study drug-1 year
The incidence of infections other than acute serious bacterial infections | during treatment with study drug-1 year
The number of days lost from work/school/usual activities | during treatment with study drug-1 year
The number of days of antibiotic therapy (prophylactic and treatment) | during treatment with study drug-1 year
Pharmacokinetic parameters of IgG subclasses and specific antibodies will be determined in at least 20 patients: AUC0-t, Cmax, Tmax, t1/2, Vd and elimination rate constants. | after 5th or 6th study infusion
Trough levels of IgG subclasses and specific antibodies will be estimated for each subject in the pharmacokinetic study at defined intervals. | Months 0, 5, 9, 12
The number of patients whose trough IgG levels fall below the target of 500 mg/dL at any time will be recorded. | one year
All adverse events that occur during the study regardless of the investigator's assessment of the relationship to the investigational product. | one year
Laboratory assessments on blood and urine samples including direct antiglobulin (Coomb's) tests. | one year
Markers of blood borne virus infections at baseline and up to 3 months after the last infusion i.e. HIV (serology), HCV (serology and NAT), HBV (HbsAg). | Months -1, 14, 16

CONTACTS AND LOCATIONS:
Overall Officials: Chaim Roifman, MD, Study Chair — The Hospital for Sick Children; Robert Roberts, MD, Principal Investigator — Mattel Children's Hospital of UCLA; Isaac R Melamed, MD, Principal Investigator — 1st Allergey and Clinical Research Center; James Moy, MD, Principal Investigator — Rush Universitity Medical Centre; Eyal Grunebaum, MD, Principal Investigator — The Hospital for Sick Children; Gordan L Sussman, MD, Principal Investigator — University of Toronto; Akhilesh Chouksey, MD, Principal Investigator — Rainbow Babies and Children's Hospital; Mark Stein, MD, Principal Investigator — Allergy Associates of the Palm Beaches; Richard L Wasserman, MD, Principal Investigator; Daniel Suez, MD, Principal Investigator — Allergy, Asthma and Immunology Clinic PA; Don McNeil, MD, Principal Investigator — Optimed Research LLC
Locations (10):
- United States (8):
  - Mattel Children's Hospital of UCLA, Los Angeles, California
  - 1st Allergy and Clinical Research Center, Centennial, Colorado
  - Allergy Associates of the Palm Beaches, North Palm Beach, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Optimed Research, LLC, Columbus, Ohio
  - Pediatric Allergy Immunology Associates, Dallas, Texas
  - Allergy, Asthma and Immunology Clinic PA, Irving, Texas
- Canada (2):
  - University of Toronto, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Background] Ten RM. Primary immunodeficiencies. Mayo Clin Proc. 1998 Sep;73(9):865-72. doi: 10.4065/73.9.865. PMID 9737224
- [Background] Bonilla FA, Geha RS. 12. Primary immunodeficiency diseases. J Allergy Clin Immunol. 2003 Feb;111(2 Suppl):S571-81. doi: 10.1067/mai.2003.86. PMID 12592303
- [Background] Bonilla FA, Bernstein IL, Khan DA, Ballas ZK, Chinen J, Frank MM, Kobrynski LJ, Levinson AI, Mazer B, Nelson RP Jr, Orange JS, Routes JM, Shearer WT, Sorensen RU; American Academy of Allergy, Asthma and Immunology; American College of Allergy, Asthma and Immunology; Joint Council of Allergy, Asthma and Immunology. Practice parameter for the diagnosis and management of primary immunodeficiency. Ann Allergy Asthma Immunol. 2005 May;94(5 Suppl 1):S1-63. doi: 10.1016/s1081-1206(10)61142-8. No abstract available. PMID 15945566
- [Background] Chapel HM. Consensus on diagnosis and management of primary antibody deficiencies. Consensus Panel for the Diagnosis and Management of Primary Antibody Deficiencies. BMJ. 1994 Feb 26;308(6928):581-5. doi: 10.1136/bmj.308.6928.581. No abstract available. PMID 8148684
- [Background] Roifman CM, Levison H, Gelfand EW. High-dose versus low-dose intravenous immunoglobulin in hypogammaglobulinaemia and chronic lung disease. Lancet. 1987 May 9;1(8541):1075-7. doi: 10.1016/s0140-6736(87)90494-6. PMID 2883406
- [Background] Eijkhout HW, van Der Meer JW, Kallenberg CG, Weening RS, van Dissel JT, Sanders LA, Strengers PF, Nienhuis H, Schellekens PT; Inter-University Working Party for the Study of Immune Deficiencies. The effect of two different dosages of intravenous immunoglobulin on the incidence of recurrent infections in patients with primary hypogammaglobulinemia. A randomized, double-blind, multicenter crossover trial. Ann Intern Med. 2001 Aug 7;135(3):165-74. doi: 10.7326/0003-4819-135-3-200108070-00008. PMID 11487483
- [Background] Roifman CM, Schroeder H, Berger M, Sorensen R, Ballow M, Buckley RH, Gewurz A, Korenblat P, Sussman G, Lemm G. Comparison of the efficacy of IGIV-C, 10% (caprylate/chromatography) and IGIV-SD, 10% as replacement therapy in primary immune deficiency. A randomized double-blind trial. Int Immunopharmacol. 2003 Sep;3(9):1325-33. doi: 10.1016/s1567-5769(03)00134-6. PMID 12890430
- [Background] Berger M. A history of immune globulin therapy, from the Harvard crash program to monoclonal antibodies. Curr Allergy Asthma Rep. 2002 Sep;2(5):368-78. doi: 10.1007/s11882-002-0069-z. PMID 12165202